CLINICAL TRIAL: NCT03766256
Title: Pilot Study of Pharmacist-Coordinated Implementation of the Diabetes Prevention Program (DPP) for Women With a History of Gestational Diabetes Mellitus (GDM)
Brief Title: Shared Decision Making in Diabetes Prevention for Women With a History of GDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Kenrik Duru, Professor of Medicine, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB#18-001058
Record Dates: First submitted 2018-11-05; First posted 2018-12-06 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Pharmacists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shared decision-making with pharmacists (Experimental): Pharmacist-coordinated shared decision making about treatment for history of gestational diabetes mellitus (lifestyle change and/or metformin), using a decision tool
  Interventions: Behavioral: Shared decision-making with pharmacists

INTERVENTIONS:
Behavioral: Shared decision-making with pharmacists — Pharmacist will engage patient with history of gestational diabetes mellitus using Healthwise (TM) Decision Tool to help match their personal preferences and values with treatment options, specifically lifestyle change will be referred to a CDC (Center for Disease Control and Prevention) approved diabetes prevention program, and pharmacists will coordinate with primary care providers to prescribe metformin for patients interested in this treatment.

SUMMARY:
Gestational diabetes mellitus (GDM) is a risk factor for the development of Type 2 diabetes. Lifestyle change and metformin are equally effective in preventing diabetes in patients with a history of GDM, so these women should choose a strategy based on their preferences and values, which may vary by race/ethnicity. This proposal will engage 32 women in shared decision making about diabetes prevention.

DETAILED DESCRIPTION:
The Diabetes Prevention Program (DPP) demonstrated that intensive lifestyle change and metformin both prevent or delay Type 2 diabetes (T2DM), but uptake of either approach has been minimal. The research team is implementing a shared decision-making (SDM) intervention for diabetes prevention funded by the National Institute of Diabetes and Digestive and Kidney Disease (NIDDK; R18 DK105464). In this clinic-based pragmatic trial, the Prediabetes Informed Decisions and Education (PRIDE) study, pharmacists engage patients with prediabetes in evidence-based diabetes prevention using an SDM framework. The research team reached the recruitment goal (n=350) more than 15 months ahead of schedule and enrolled 1.5 times the number of projected participants (n=515), including 56% from racial/ethnic minority groups. PRIDE has been highly successful in treatment engagement, as 85% of participants chose either lifestyle change or metformin. Furthermore, among patients who have reached 12-month follow-up, PRIDE participants as a group have lost more weight than matched controls (-5.2 lbs. vs. -0.29 lbs., p<0.001).

PRIDE targets both men and women with prediabetes. Only five PRIDE participants had a history of gestational diabetes mellitus (GDM) during a prior pregnancy. GDM is more common among minority women and a history of a GDM diagnosis is one of the most significant risk factors for incident type 2 diabetes, increasing the risk of developing T2DM upwards of sevenfold. The research team is planning to pilot an SDM intervention for women with a history of GDM. This project would advance a patient-centered approach to increase uptake of both evidence-based diabetes prevention strategies among the subgroup of minority women at the highest risk of progression to T2DM.

In the proposed project, the research team plans to enroll women with a history of GDM in a pilot study, tracking their choice of diabetes prevention strategy and their weight change over time. Importantly, the pilot will enable the research team to estimate the sample size for a future, multi-center study to engage women with a history of GDM in SDM for diabetes prevention. The project's specific aim is as follows:

In a pilot study, to deliver the tailored intervention to a diverse sample of 32 women with a history of GDM and hemoglobin A1c from 5.7-6.4% who have not yet developed Type 2 diabetes, with a sample divided equally between whites, African Americans, Latinas and Asian Americans

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese (BMI >25 or >23 if Asian American)
* at least 6 weeks post-partum
* have a history of gestational diabetes mellitus

Exclusion Criteria:

* Currently pregnant,
* not a UCLA Health patient
* any history of a Type 2 diabetes diagnosis, based on billing codes, laboratory values, or taking any antiglycemic medications

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 33 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Choice of evidence-based diabetes prevention (lifestyle change or metformin) | 2 weeks
  One of four participant decisions: 1) choosing to attend a Centers for Disease Control and Prevention (CDC)-certified diabetes prevention program, 2) choosing to start metformin as diabetes prevention, 3) choosing both the diabetes prevention program and metformin, 4) choosing NOT to start either the diabetes prevention program or start metformin.

SECONDARY OUTCOMES:
Weight change | 9 months
  Change of weight as measured in the EHR
Systolic blood pressure | 9 months
  Change in systolic blood pressure as measured in the EHR
Decisional conflict | 2 weeks
  Three collaboRATE items that measure decisional conflict

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Toluca Lake Health Center, Burbank, California
  - 100 Medical Plaza Primary Care Suites 455 & 490, Los Angeles, California
  - Internal Medicine Women's Health Clinic Suites 250 & 290, Los Angeles, California
  - UCLA Internal Medicine Family Westwood Suite 465, Los Angeles, California
  - UCLA Internal Medicine Geriatrics Suite 365 & 420, Los Angeles, California
  - CPN Brentwood, Los Angeles, California
  - CPN West Washington Internal Medicine, Los Angeles, California
  - Pacific Palisades, Pacific Palisades, California
  - 12th Street Clinic, Santa Monica, California
  - Wilshire Office, Santa Monica, California
  - CPN Santa Monica 15th Street Family Medicine Practice, Santa Monica, California
  - CPN/Santa Monica Parkside, Santa Monica, California
  - Santa Moica Bay Physicians/20th Street 10th Floor, Santa Monica, California
  - Santa Monica Bay Physicians Plaza, Santa Monica, California
  - Santa Monica Bay Physicians/20th Street 3rd Floor, Santa Monica, California
  - Santa Monica Internal Medicine, Santa Monica, California
  - UCLA Family Health Clinic, Santa Monica, California
  - Santa Moica Bay Physicians Ocean Park, Santa Monica, California
  - Jack H. Skirball Health Center, Woodland Hills, California
  - CPN Woodland Hills Practice, Woodland Hills, California

REFERENCES:
- [Derived] Madievsky R, Vu A, Cheng F, Chon J, Turk N, Krueger A, Krong J, Maranon R, Liu S, Han CS, Norris KC, Mangione C, Page J, Thomas S, Duru OK, Moin T. A randomized controlled trial of a shared decision making intervention for diabetes prevention for women with a history of gestational diabetes mellitus: The Gestational diabetes Risk Attenuation for New Diabetes (GRAND study). Contemp Clin Trials. 2023 Jan;124:107007. doi: 10.1016/j.cct.2022.107007. Epub 2022 Nov 13. PMID 36384219